CLINICAL TRIAL: NCT01604317
Title: Randomized Evaluation of the Use of Plastic Bags to Prevent Neonatal Hypothermia in Developing Countries-Part I
Brief Title: Evaluation of Use of Plastic Bags to Prevent Neonatal Hypothermia-Part I
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Children's Health System, Alabama (Other)
Responsible Party: Principal Investigator, Waldemar A. Carlo, Edwin M. Dixon Professor of Pediatrics, Director of Division of Neonatology, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UAB Neo 005; Perinatal Health/Human (Other: University of Alabama at Birmingham); Childrens Centennial (Other: Childrens of Alabama); Caduceus Club (Other: University of Alabama School of Medicin)
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Hypothermia; Immature Newborn
Keywords: Hypothermia; Low birth Weight; Newborn; Resuscitation; Plastic bag
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resuscitation-torso plastic bag (Active Comparator): Resuscitation with plastic bag covering torso and lower extremities for first hour to assist with temperature regulation.
  Interventions: Procedure: Resuscitation-torso plastic bag
- Resuscitation-partial-head plastic bag (Active Comparator): Resuscitation with plastic bag covering torso, upper and lower extremities, and a portion of the head for first hour after birth to assist with temperature regulation.
  Interventions: Procedure: Resuscitation-partial-head plastic bag

INTERVENTIONS:
Procedure: Resuscitation-torso plastic bag — Infant's extremities and torso will be placed in a plastic bag during resuscitation after birth and maintained for 1 hour after birth.
  Arms: Resuscitation-torso plastic bag
Procedure: Resuscitation-partial-head plastic bag — Infant's torso, extremities, and portion of the head (face will be exposed) will be placed in a plastic bag during resuscitation after birth and maintained for 1 hour after birth.
  Arms: Resuscitation-partial-head plastic bag

SUMMARY:
The overall hypothesis is that plastic bags used in combination with WHO thermoregulation care will reduce the incidence of hypothermia in preterm/low birth weight and full term infants when compared to routine WHO thermoregulation care alone. Part I is for preterm/low birth weight infant with or without plastic head cover used during resuscitation.

DETAILED DESCRIPTION:
This study will compare the incidence of hypothermia during the first hour after birth in preterm/low birth weight infants randomized to receive WHO thermoregulation care and a plastic bag (without drying) covering the torso and lower extremities (control group) or WHO thermoregulation care and a plastic bag (without drying) covering the torso, upper and lower extremities, and a portion of their head (intervention group). The axillary temperature of each infant will be taken initially within 15 minutes of birth and later at 1 hour after birth as the infant is removed from the plastic bag. Seizures, hyperthermia, room temperature, and death will be recorded throughout the hospitalization for all infants. With an estimated baseline hypothermia rate of 41% and a 21% absolute risk reduction (51% relative risk reduction), a sample size of 182 will be used to have a power of 80% and a confidence interval of 95%.

ELIGIBILITY:
Inclusion Criteria:

* Estimated gestational age 29-36 6/7weeks or birth weight 1,400-2500g
* Delivery in the hospital

Exclusion Criteria:

* Infant admitted to the NICU
* Birth weight less than 1,400g
* Abdominal wall defect or myelomeningocele
* Major congenital anomalies
* Blistering skin disorder

Ages: 1 Minute to 1 Hour | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 182 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Axillary temperature < 36.5 degrees Celsius | 1-72 hours after birth
  Temperature taken per axilla at one hour after birth. Temperatures 36.0-36.4 will be classified as mild hypothermia, 32.0-35.9 will be classified as moderate hypothermia, and < 32.0 will be classified as severe hypothermia

SECONDARY OUTCOMES:
Seizure | Up to 4 weeks
  Seizure activity diagnosed by medical doctor or nurse. No electroencephalogram will be done.
Respiratory Distress Syndrome (RDS) | Up to 4 weeks
  Documentation of increased work of breathing, retractions, and a need for oxygen, intubation, or surfactant
Pneumothorax | Up to 4 weeks
  Either chest radiograph documentation or clinical deterioration consistent with air leak
Sepsis | Up to 4 weeks
  Culture proven or culture negative clinically treated course consistent with sepsis
Necrotizing enterocolitis or intestinal perforation | Up to 4 weeks
  Documentation of pneumatosis or intestinal perforation on x-ray or treatment course for clinical necrotizing enterocolitis per Bell's classification stage greater than one.
Death | Up to 4 weeks
  Cardiorespiratory failure
Hyperthermia | Up to 4 weeks
  Axillary temperature > 38 degrees Celsius per temperature taken per axilla for one minute
Temperature and humidity | 1-72 hours after birth
  A recording of the room temperature and humidity will be obtained with each axillary temperature measurement

CONTACTS AND LOCATIONS:
Overall Officials: Waldemar A Carlo, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University Teaching Hospital, Lusaka, Zambia